CLINICAL TRIAL: NCT03171246
Title: An Open Label Pilot Study of the CD-TREAT Diet as a Novel Therapy for Active Luminal Crohn's Disease
Brief Title: CD-TREAT Diet: a Novel Therapy for Active Luminal Crohn's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GN17GA213P
Record Dates: First submitted 2017-05-17; First posted 2017-05-31 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Crohn Disease
Keywords: dietary intervention
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD-TREAT (Solid food-based intervention) (Experimental): Solid food-based dietary intervention replicating composition of exclusive enteral nutrition (EEN).
  Daily for up to 12 weeks.
  Interventions: Dietary Supplement: Solid food-based intervention

INTERVENTIONS:
Dietary Supplement: Solid food-based intervention — Individually tailored energy content according to age/activity

SUMMARY:
Crohn's disease (CD) is a chronic inflammatory condition of the gut with severe complications. There is strong evidence to suggest that diet and gut bacteria are key components in the onset, perpetuation and management of CD.

An 8-week exclusive liquid diet (EEN) without any normal food is the best treatment for paediatric CD. The mode of action of EEN remains unknown, but according to recent publications, the modulation of the gut bacteria drives its therapeutic properties. While successful, EEN is a challenging therapy to follow. Half of the paediatric EEN patients will require a nasogastric tube to support treatment, its use in adults is limited, and the need for a more palatable diet is very well described. Based on these findings, a non-liquid and more acceptable dietary treatment was recently devised called CD-TREAT (Crohn's Disease TReatment-with-EATing) diet. CD-TREAT, which is a solid food-based diet designed to replicate the nutrients and food ingredients composition of EEN, was recently tested in healthy adults and a rat model of colitis. In order to pilot CD-TREAT diet as a CD induction treatment, 10 children and 10 adults with active luminal CD will be recruited. Once consented, baseline blood, urine and faecal samples will be collected and the CD-TREAT prescribed for a maximum of 12 weeks. Another 3 blood, urine and faecal samples will be requested during the 12 weeks. All the foods/meals of the CD-TREAT diet will be purchased and delivered to the participants' house by the researcher and the meals which need cooking will be pre-prepared by a sub-contracted catering company. Blood and faecal inflammatory biomarkers will be measured, the disease activity assessed with routinely used clinical indices and the faecal bacteria and its metabolites characterised.

DETAILED DESCRIPTION:
Children and adults who are eligible to participate will be identified by medical staff. A member of the clinical team will briefly inform potential participants about the study via the phone, via e-mail, or at the clinic. After the end of the clinical appointment and if the patient and/or the parent/carer are agreeable, a member of the clinical team will introduce the eligible participants to the researcher who will explain the study in full and answer any questions they might have. During this meeting, the researcher will discuss the specific aspects of dietary treatment with CD-TREAT and will inform participants that urine, blood and faecal samples will be collected to try and determine the type of bacteria which may be associated with gut inflammation, and their metabolites, and whether these can predict response to treatment. The researcher will also ask for permission to collect medical information from the participant's medical records. If they are interested in taking part, they will be given detailed written information (including an age-appropriate information leaflet). The information pack will also invite the family to contact the researcher at any time if they require further information.

As there is a very narrow time window between identification of eligible participants and consent to participate to the study, and considering the need for immediate initiation of treatment in patients with active disease, it is anticipated that signed consent to join the study will be obtained on the same day of receiving information about it; however there will be subsequent opportunity to review this decision. Consent will only be taken if participants feel they have had adequate time to make this decision, and no pressure will be applied in any way.

This will also facilitate the completion of a health check questionnaire, baseline clinical review, medication and disease history, quality of life assessment, anthropometry measurements, collection of baseline research bloods (extra volume at the time of routine clinical tests (no additional venepuncture required). At this point the participant will be asked to take a stool and urine sample collection kit at home and a suitable date/time to collect the baseline samples will be arranged. The actual intervention will start approximately 24 hours later in order to allow the participants enough time to consider and discuss the study with their relatives, decide whether they would like to continue or drop out and start the standard induction treatment as deemed necessary by the treating clinical team. Furthermore, this 24 hour time window will enable the researcher to collect baseline samples before the initiation of the CD-TREAT dietary treatment.

Where appropriate, the assent of the child will be sought (usually under age 11 or younger), and in the case of young adults who would be deemed able by a member of the clinical team to consent on their own part (usually age 12 or older), consent from the young person will be accompanied by the parent/carer giving signed assent before they can join the study; to ensure both child and parent/carer are willing and happy to take part. For children unable to give written consent/assent, the parent/carer will be asked to explain the study in terms that the child can understand and the carer will sign consent on their behalf.

It will also be made clear at this stage, on information sheets and throughout the study that participants can withdraw from the study at any time without it affecting their routine care in any way. Continuation of CD-TREAT dietary advice and provision of CD-TREAT foodstuffs is dependent however on continuation in the study. Discontinuation of study participation after commencement of CD-TREAT would therefore involve return to standard induction treatment at the discretion of the treating clinical team.

Throughout the study recruited participants will be asked to provide urine, faecal and blood samples (an additional small tube of blood when they are having routine bloods at clinical appointments) on a maximum of 4 occasions. In addition, these time points will include clinical review, quality of life assessment and anthropometry measurements.

Participants will also provide some dietary information reflecting their compliance to CD-TREAT diet.

CD-TREAT Intervention:

All patients on the CD-TREAT diet will be supplied with an individually tailored, dietitian-devised diet, consisting of ordinary foods, but custom-designed to recreate the nutritional content and ingredients of EEN. The dietary intervention will be overseen by qualified dieticians including a National Health Service (NHS) research dietician. The energy content will be tailored to adult participants' total energy expenditure and physical activity level calculated by the World Health Organisation (WHO) set of equations or will be calculated for each child to meet their estimated average requirement (EAR) for age. Food and instructions for those patients on CD-TREAT will be supplied directly to them by the researchers on the day following recruitment. Foods which need cooking will be prepared by a sub-contracted (food handling and hygiene certified) catering company and will be delivered to the participants' house every 2-3 days. The rest of the foods will be delivered to the participants' house every week. Participants will initially receive the modified diet for a period of 8 weeks, similar to the duration of an EEN course. The researchers will instruct the participants and their carers on how to follow the diet and how to record their dietary intake during the intervention. Research follow-up visits will coincide with the participants' clinical follow-ups (Week 2: phone review; Weeks 4 & 8: hospital visit). These follow up appointments will include collection of research bloods as an extra aliquot to their routine clinical tests (no additional needle insertion is required), clinical review, quality of life assessment and anthropometry measurements. At these appointments, the researchers will give the participants a stool and urine sample collection kit to take home and will arrange a suitable date/time to collect the faecal and urine sample.

Response to treatment will be assessed according to clinical review, CD activity score and measurements of established biomarkers in faeces and blood (e.g. faecal calprotectin). The primary endpoint will be clinical response (Adults: HBI fall≥3; Children: wPCDAI fall≥17.5) or clinical remission (Adults: HBI<5; Children: wPCDAI<12.5) at 8 weeks; while secondary endpoints include reduction in faecal calprotectin and blood inflammatory markers and changes in anthropometry. All patients will be under close follow-up. No new CD-related medications will be allowed during the pilot study, however if patients' disease activity is deteriorating at any point during the study or there is no response at 4 weeks, patients will be eligible to discontinue CD-TREAT diet and commence medical/surgical treatment as deemed necessary by the treating clinical team. Those participants will still be encouraged to provide stool, blood and urine samples at intervention exit. For those demonstrating response, all background CD-related medication dosages will remain stable unless a subject develops specific drug-related side-effects, blood monitoring abnormalities or blood drug levels requiring alteration. Those patients who experience clinical response but not clinical remission at 8 weeks will be given the opportunity to stay on CD-TREAT for a further 4 weeks. At the end of this period (12 weeks post CD-TREAT initiation) they will be asked to provide the last stool and urine sample and they will have the last follow-up appointment including collection of research bloods, clinical review, quality of life assessment and anthropometry measurements.

ELIGIBILITY:
Inclusion Criteria:

* previously diagnosed patients with active luminal CD [paediatric (6-15 years old) wPCDAI≥12.5) or adult (16-65 years old) HBI≥5]
* in need of starting induction treatment

Exclusion Criteria:

* pregnancy
* use of antibiotics currently or during the past 1 month
* major change in inflammatory bowel disease (IBD) induction or maintenance therapy in the preceding 3 months (defined as change in type of treatment)
* minor change in IBD induction or maintenance therapy in the preceding 1 month (defined as adjustment of treatment dosage)
* enrolment in other studies investigating the efficacy of other novel therapies in disease activity
* disease severity sufficient to warrant hospital admission
* food allergies incompatible with CD-TREAT (e.g. cow's milk allergy)

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Crohn's Disease activity | Baseline to 8 weeks
  Change in Harvey Bradshaw Index (HBI) (adults) or weighed Paediatric Crohn's Disease Activity Index (wPCDAI) (children) score

SECONDARY OUTCOMES:
Faecal calprotectin | Baseline to 8 weeks
  Change in faecal calprotectin level
Blood inflammatory marker | Baseline to 8 weeks
  Change in blood inflammatory marker level
Height | Baseline to 8 weeks
  Change in height (cm)
Quality of Life | Baseline to 8 weeks
  Change in Self-Administered Inflammatory Bowel Disease Questionnaire (SIBDQ) (adults) and IMPACT III (children) score
Weight | Baseline to 8 weeks
  Change in weight (kg)
Body Mass Index | Baseline to 8 weeks
  Change in Body Mass Index (BMI)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Hansen, MB ChB MRCPCH PhD, Principal Investigator — NHS Greater Glasgow and Clyde
Locations (2):
- United Kingdom (2):
  - Glasgow Royal Infirmary, Glasgow, Scotland
  - Royal Hospital for Children, Glasgow, Scotland

IPD SHARING:
Plan to Share IPD: Yes
Participants will be asked to provide written consent for their anonymised data to be made available to public data repositories.

REFERENCES:
- [Derived] Svolos V, Hansen R, Nichols B, Quince C, Ijaz UZ, Papadopoulou RT, Edwards CA, Watson D, Alghamdi A, Brejnrod A, Ansalone C, Duncan H, Gervais L, Tayler R, Salmond J, Bolognini D, Klopfleisch R, Gaya DR, Milling S, Russell RK, Gerasimidis K. Treatment of Active Crohn's Disease With an Ordinary Food-based Diet That Replicates Exclusive Enteral Nutrition. Gastroenterology. 2019 Apr;156(5):1354-1367.e6. doi: 10.1053/j.gastro.2018.12.002. Epub 2018 Dec 11. PMID 30550821